CLINICAL TRIAL: NCT00917176
Title: Subcutaneous C2 Stimulation: Treatment of Fibromyalgia
Brief Title: Occipital Nerve Stimulation in Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof. Dr. Dirk De Ridder, University Hospital Antwerp
Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMS_ONS_01
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Effective stimulation (Experimental): Effective stimulation at sub-threshold level
  Interventions: Device: Occipital nerve stimulation
- Placebo stimulation (Placebo Comparator): Stimulation at non-effective strength
  Interventions: Device: Occipital nerve stimulation

INTERVENTIONS:
Device: Occipital nerve stimulation

SUMMARY:
The aim of this study is to investigate whether greater occipital nerve stimulation is effective in the treatment of fibromyalgia related pain. The study uses sub sensory threshold stimulation and placebo stimulation in order to investigate whether sub-threshold stimulation is feasible in a placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed according to the criteria of the American College of Rheumatology (ACR-90)
* Minimally treated with adequate trials during 3 months
* Insight of the patient in her disease and capable of understanding and signing an informed consent

Exclusion Criteria:

* History of severe illness or suffering from severe chronic disease
* History of substance abuse, unless treated and in remission during 6 months
* Cardiac disease
* History of epileptic insults
* Psychiatric disorders with psychotic symptoms
* Pace maker / defibrillator
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Pain scores on Visual Analogue Scale (VAS), pain Catastrophizing Scale (PCS), pain vigilance and awareness questionnaire (PVAQ) | at a weekly base during 10 weeks

SECONDARY OUTCOMES:
Scores on Fatigue and Mood | at a weekly base, during 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ridder, M.D., PhD., Study Chair — University Hospital, Antwerp; Mark Plazier, M.D., Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Belgium

REFERENCES:
- [Derived] Ahmed S, Plazier M, Ost J, Stassijns G, Deleye S, Ceyssens S, Dupont P, Stroobants S, Staelens S, De Ridder D, Vanneste S. The effect of occipital nerve field stimulation on the descending pain pathway in patients with fibromyalgia: a water PET and EEG imaging study. BMC Neurol. 2018 Nov 12;18(1):191. doi: 10.1186/s12883-018-1190-5. PMID 30419855